CLINICAL TRIAL: NCT02766426
Title: Cytokine and Body Composition's Changes Throughout Pregnancy in Overweight/Obese Women Undergoing an Early Lifestyle Change Program
Brief Title: Cytokine and Body Composition's Changes in Overweight/Obese Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Prof. Facchinetti Fabio, Chairman of Obstetrics and Gynecology Unit, University of Modena and Reggio Emilia
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 136/15
Record Dates: First submitted 2016-04-14; First posted 2016-05-09 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-04

CONDITIONS: Maternal Obesity Complicating Pregnancy; Exercise Addiction; High-Risk Pregnancy; Inflammatory Status During Preganancy; Maternal Body Composition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lifestyle change intervention (Other): Overweight/obese pregnant women enrolled in a healthy lifestyle change programm
  Interventions: Behavioral: Lifestyle change program

INTERVENTIONS:
Behavioral: Lifestyle change program — Women attended a multidisciplinary counseling (by both the dietitian and the gynecologist). They were given nutritional advice about lifestyle and physical activity, in agreement with the Italian Guidelines for a healthy diet during pregnancy. The diet given comprised 1500 kcal/day and consisted of 3 main meals and 3 snacks (breakfast, snack, lunch, snack, dinner, and evening snack) that corresponds to the baseline metabolism of a pregnant woman. In view of the physical activity program, the dietitian added an amount of 200 kcal/day for obese or 300 kcal/day for overweight women.
  The exercise intervention was focused on increasing walking and developing a more active lifestyle. The recommendation for physical activity was to perform 30 min of moderate intensity activity at least 3 days a week.

SUMMARY:
Sincev the adipose tissue as been identified as a metabolic active tissue that produces and regulates pro-inflammatory factors, the investigators studied the relationship between cytokine changes and maternal body composition.

The investigators evaluated plasmatic pro- and anti-inflammatory cytokines levels in pregnant women with BMI >25 Kg/m^2 undergoing a lifestyle change program, and if this is related with changes in body composition.

Women enrolled in the study were provided nutritional advices about lifestyle: a proper nutrition and a constant physical activity (30 minutes/day, 3 times/week, according to the American College of Obstetricians and Gynecologists Guidelines) in an integrated counselling with a dietitian and a gynaecologist, both attendant since the enrollment.

Plasma pro- and anti-inflammatory markers were investigated at enrollment (9-12 weeks) and at 36-38 weeks.

Furthermore, the investigators used the bioimpedance analyzer to evaluate changes of body composition (i.e. fat mass and fat free mass) at first and third trimester.

DETAILED DESCRIPTION:
Pregnant women, recruited from antenatal clinics, with pre-pregnancy BMI ≥ 25 kg/m2, age >18 years and singleton pregnancy were enrolled within 12th week at the Obstetric Unit of Policlinico Hospital of Modena.

Exclusion criteria were as follows: twin pregnancies, chronic diseases (i.e., diabetes mellitus, chronic hypertension, untreated thyroid diseases) and dietary supplements or herbal products known to affect body weight, other medical conditions that might affect body weight.

At the first visit, an accurate obstetric history, family history, and personal history was collected for the assessment of exclusion criteria. The blood pressure, height and weight were measured, and the BMI is calculated.

Eligible women were given nutritional advices about lifestyle and physical activity, in agreement with the Italian Guidelines for a healthy diet during pregnancy. The diet given comprised 1500 kcal/day and consisted of 3 main meals and 3 snacks (breakfast, snack, lunch, snack, dinner, and evening snack) that corresponds to the baseline metabolism of a pregnant woman. In view of the physical activity program, the dietitian added an amount of 200 kcal/day for obese or 300 kcal/day for overweight women.

The exercise intervention was focused on increasing walking and developing a more active lifestyle (i.e., walking rather than driving for short distances). The recommended exercise prescription for pregnant women was generally consistent with recommendations for the general adult population. All participants were advised to participate in 30 min of moderate intensity activity at least 3 days a week.

Each subject taking part at the study received a 75-g 2-h Oral Glucose Tolerance Test (OGTT) at 16-18 and/or 24-28 weeks. The diagnosis of gestational diabetes mellitus was made for any glucose value exceeding the normal cut-off, as reported by the Guidelines. If OGTT is pathological, women are referred to other health care specialists for further clinical evaluation and/or specific treatment.

Women were scheduled to have a specific follow-up visits for adherence to the program at 16th, 20th, 28th and 36th week also evaluating the fat mass, fat-free mass and total body water through the use of the bioimpedance analyzer.

Furthermore, at baseline and at 36-38 week, blood plasma samples were collected in order to investigate: plasma pro- and anti-inflammatory markers related to obesity and to visceral adipose tissue (interferon-γ, interleukin-1α, interleukin-1β, interleukin-2, interleukin-4, interleukin-6, interleukin-8, interleukin-10, interleukin-12p70, and tumor necrosis factor-α).

Data regarding pregnancy and delivery were collected from clinical diaries.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* single pregnancy

Exclusion Criteria:

* twin pregnancies
* chronic diseases (i.e., diabetes mellitus, chronic hypertension, untreated thyroid diseases)
* dietary supplements or herbal products known to affect body weight
* other medical conditions that might affect body weight

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-04 (Actual); Study Completion 2016-05

PRIMARY OUTCOMES:
Cytokine changes throughout pregnancy in overweight/obese women undergoing a lifestyle change program. | At baseline, at 36-38 week
  interferon(IFN)-γ, interleukin(IL)-1α, IL-1β, IL-2, IL-4, IL-6, IL-8, IL-10, IL-12p70, and tumor necrosis factor-α plasma levels (pg/ml)
Weight changes | At baseline, at 36 weeks
  Weight at baseline (i.e. enrollment: 9 weeks) and at 36 weeks measured in kg
Fat mass changes | At baseline, at 36 weeks
  Changes in total and visceral (trunk) fat mass (FM) at baseline (i.e. enrollment: 9 weeks), at 36 weeks and calculated as fat changes

CONTACTS AND LOCATIONS:
Locations (1):
- Mother-Infant Department, University of Modena and Reggio Emilia, Italy, Modena, Italy

IPD SHARING:
Plan to Share IPD: No